CLINICAL TRIAL: NCT04194333
Title: Comparing Diagnostic Yield of Electromagnetic Navigational Bronchoscopy Guided With Real Time Cone Beam Computer Tomography With Standard Fluoroscopy Guidance for Peripheral and Central Lung Lesions
Brief Title: Cone Beam CT Guided Electromagnetic Navigational Bronchoscopy
Acronym: CBCTENB
Status: Completed | Type: Observational
Sponsor: Columbus Regional Health (Other)
Responsible Party: Principal Investigator, Deepankar Sharma, Medical Director, Lung Institute and Section Chief, Pulmonary & Critical Care, Columbus Regional Health
Other Study IDs: 001
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Lung Nodule; Lung Mass; Lesion of the Lung
Keywords: Lung Nodule; Lung Mass; Lung Lesion; Cone Beam CT; CT Augmented Fluoroscopy; EMN; Electromagnetic Navigation Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Fluoroscopy Guided EMN: Patient is undergoing electromagnetic navigation bronchoscopy using Medtronic super D version 7 EMN system, peripheral endobronchial ultrasound and standard fluoroscopy using the C-arm under general anesthesia.
- Cone Beam CT Guided EMN: Patient is undergoing electromagnetic navigation bronchoscopy using Medtronic super D version 7 EMN system, peripheral endobronchial ultrasound and Cone Beam CT Guidance using the Philips Azurion 7 C20 FlexMove with Embo Guide and Overlay software to create CT Augmented Fluoroscopy under general anesthesia.
  Interventions: Procedure: Cone Beam CT with Embo Guide to creat 3D Overlay and CT Augmented Fluoroscopy to guide Electromagnetic Navigational Bronchoscopy instead of Standard Fluroscopic guidance using the C-Arm

INTERVENTIONS:
Procedure: Cone Beam CT with Embo Guide to creat 3D Overlay and CT Augmented Fluoroscopy to guide Electromagnetic Navigational Bronchoscopy instead of Standard Fluroscopic guidance using the C-Arm — Instead of the standard fluoroscopy using the C-arm, the intervention will undergo electromagnetic navigation guided bronchoscopy while using Cone Beam CT with Embo Guide to creat 3D Overlay and CT Augmented Fluoroscopy.
  Groups: Cone Beam CT Guided EMN

SUMMARY:
Electromagnetic navigation bronchoscopy (ENB) is used to access peripheral and central parenchymal lung lesions via endobronchial and transbronchial approach. Traditionally ENB is done under fluoroscopic guidance using C-arm but with development of Cone Beam CT and 3D reconstruction technology, fluoroscopy can be enhanced to much higher resolution and can also provide real time 3D augmentation of the lesion. It also enables the user to obtain a CT of the Chest to confirm the real time location of the lesion and the bronchoscopic biopsy catheter and instruments. This is thought to improve the yield and sensitivity of ENB guided Biopsy of the lung nodules and masses but has not been proven in a prospective trial. With my study, I want to examine the effect of Cone Beam CT with 3D reconstruction on the diagnostic yield and sensitivity of Electromagnetic Navigational Bronchoscopic biopsy of the lung lesions.

DETAILED DESCRIPTION:
Electromagnetic navigation bronchoscopy has been used for more than a decade to access peripheral and central parenchymal lung lesions bronchoscopically. Traditionally standard fluoroscopy using C-arm is used to confirm the location and guide the biopsy instruments under real-time guidance. With availability of Cone Beam CT, fluoroscopic images of much higher quality and resolution can be obtained intra-operatively. It also enables the bronchoscopist to obtain intraoperative CT images and confirm the exact location of the lesion and the Bronchoscopic biopsy catheter or the biopsy instruments.

At my institution, lung nodules/masses requiring ENB have been approached using Medtronic Super-Dimension Version 7 Electromagnetic Navigational Bronchoscopy system. All the procedures are done under fluroscopic guidance using a regular C-Arm. All the lesions are confirmed using peripheral Endobronchial Ultrasound (EBUS). Once the appropriate location is reached, biopsy is obtained using FNA (18G or 21G), Single or Triple needle brush, Transbronchial forceps and Bronchoalveolar lavage.

A pathologist is present on site for all the cases to review the slides and assist in diagnosis. All the cases are done under general anesthesia through endotracheal tube.

Also, all the ENB procedures have been performed by one Interventional Pulmonologist since August 2017.

For the interventional arm, all the aspects will remain the same except that the cases are done in Hybrid OR instead of Endoscopy. All the patients are completely paralyzed intra-operatively. Also, instead of a standard C-Arm providing 2D fluoroscopic guidance, a Philips Azurion 7 C20 FlexMove system with Emboguide, 3D Segmentaion and Overlay tools is being used. This enables the bronchoscopist to obtain a CT scan of the chest and also segment out the lesion(s) of interest and to overlap the 3-D image of the lesion on live fluoroscopy in all 3 dimensions.

During the ENB procedures, at least 1 full Xpert CT is going to be obtained, mostly after completing the airway registration and ENB guided approach the lesion. Once the extended working channel and the locatable guide is advanced to the lesion using ENB guidance, the catheter is locked and scope held in place. The patient is maintained in inspiratory breath hold and Cone Beam Ct is used to obtain the Xpert CT that shows the lesion and surrounding lungs, chest and mediastinal structures in the surrounding area of the chest.

This is then used to analyze the location of the lesion and the lesion of the extended working channel, locatable guide and the biopsy instruments in relation to the lesion. The lesion is then segmented and EmboGuide+Overlay feature is used to project a 3D view of the lesion on the live fluoroscopic images in all three axis. This also allows the bronchoscopist to obtain Anterior-posterior, Lateral and oblique views at various angles while maintaining the 3D overlap.

Additional CT scans might be obtained intra-operatively if needed to guide the biopsy catheter appropriately towards the lesion. Due to the live nature of the Cone Beam CT, it is much more capable of providing accurate guidance regarding the location of the lesion and the biopsy instruments. hence, in case of any discrepancy, information provided by Cone Beam CT is considered more reliable and used with higher confidence.

Rest of the steps involved in procedure are similar between the control and the interventional arm including the surgeon, type of bronchoscopes, type of electromagnetic navigational system, use of peripheral Endobronchial Ultrasound and availability of on-site pathologist. The biopsy instruments used are also the same including transbronchial needle for FNA, Single or triple needle brush and transbronchial forceps. Bronchoalveolar lavage is also obtained at the end via extended working channel.

All the patients undergoing biopsy of the peripheral/central lung lesions using ENB also undergo Convex EBUS guided mediastinal surveillance and EBUS-TBFNA of any Lymph Node that appears to be greater than 5 mm on EBUS exam.

My study aims to study the effect of using Cone Beam CT with segmentation, 3-D overlay and CT augmented fluoroscopy on sensitivity and diagnostic yield of electromagnetic navigation bronchoscopy for diagnosis of peripheral and central lung lesions including lung nodules and masses which could not be directly accessed using just white light bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung nodule
* Patients with lung mass
* Patients undergoing undergoing electromagnetic navigation bronchoscopy for biopsy.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients unable to complete the electromagnetic navigational bronchoscopy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodule, mass or lesion undergoing electromagnetic navigation bronchoscopy for biopsy. Majority of the patients are smokers. Some of the patients are found to have the lung nodule, mass or lesion incidentally or on the low-dose CT for lung cancer screening.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity for malignancy | 1 year Follow up. Prelim results to be reviewed at 3 months
  Percentage of malignant lesions accurately diagnosed on biopsy
Diagnostic Yield | 1 year Follow up. Prelim results to be reviewed at 3 months
  Percentage of correct underlying diagnosis

SECONDARY OUTCOMES:
Procedural Complications | 1 year Follow up. Prelim results to be reviewed at 3 months
  Pneumothorax or Bleeding
Procedure Time | 1 year Follow up. Prelim results to be reviewed at 3 months
  Intra-Operative time
Radiation Exposure | 1 year Follow up. Prelim results to be reviewed at 3 months
  Will have a record of radiation dose for the Cone Beam CT cases but not for the C-Arm cases. Will compare the radiation exposure in the Intervention arm to the average reported radiation exposure in literature.

CONTACTS AND LOCATIONS:
Overall Officials: Deepankar Sharma, MD, Principal Investigator — Columbus Regional Health
Locations (1):
- Columbus Regional Health, Columbus, Indiana, United States

IPD SHARING:
Plan to Share IPD: No